CLINICAL TRIAL: NCT03184909
Title: Consumption of Tulsi and Its Effects on Neurocognition, Stress and Anxiety: A Randomised Controlled Clinical Trial
Brief Title: Tulsi Consumption and Its Effects on Cognition, Stress and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Composite Interceptive Med Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OI-006-2017
Record Dates: First submitted 2017-06-02; First posted 2017-06-14 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Change
MeSH Terms: interventions — holy basil leaf extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Concealment of allocation and blinding of active versus placebo and blinded assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tulsi active (Experimental)
  Interventions: Drug: Ocimum Sanctum
- Tulsi placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocimum Sanctum — Active capsules containing leaves of organically prepared ocimum sanctum
  Arms: Tulsi active
Drug: Placebo — Placebo capsules of look alike inert substance for control
  Arms: Tulsi placebo

SUMMARY:
Tulsi and its effects on facilitative cognitive enhancement through lowering levels of stress and anxiety. A randomised placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Ocimum Sanctum or Holy Basil, commonly called Tulsi is a traditional Indian herb. It is believed to bring about a facilitative enhancement of cognitive ability and lower stress levels in individuals. Stress and an inability to perform at a required level of cognition can induce anxiety. This study is looking at the effects of daily consuming Tulsi among a group of individuals who work in an environment that demands memory, attention and executive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 50 years, providing written informed consent.

Exclusion Criteria:

Subjects who meet the following criteria

* Education level below 8th grade of schooling
* Unable to read or understand English or having no working knowledge of English
* Known history or neurological conditions that can affect cognition
* Known history of drug abuse or potential for drug abuse, a regular consumer of alcohol or unwilling to withhold consumption of alcohol for the duration of the study.
* A chronic smoker or consumer of other tobacco related products or is undergoing a rehabilitation program for alcohol and or tobacco consumption
* Any history or psychiatric disorders - currently on treatment or treated in within the last 12 months
* Any characteristic that makes the investigator uncomfortable to include the subject in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
To assess a change in facilitative cognitive function from baseline in 6 weeks by comparing the results on cognitive tests measured by Cambridge Neuropsychological Test Automated Battery (Cantab®) between active and placebo group | 6 weeks
  The Cambridge Neuropsychological Test Automated Battery (CANTAB) is a digital tool to measure the cognitive function.

SECONDARY OUTCOMES:
To measure change in cortisol level from saliva in 6 weeks | 6 weeks
  Salivary levels of cortisol correlates with work related stress levels. Our intention is to evaluate the effect of ocimum sanctum in lowering stress and measured as a change in the cortisol levels
To measure change in Generalized Anxiety Disorder 7-Item Scale in 6 weeks | 6 weeks
  It is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder (GAD)

CONTACTS AND LOCATIONS:
Overall Officials: Alben Sigamani, MD, Principal Investigator — Narayana Hrudayalaya Limited
Locations (1):
- Narayana Hrudayalaya Limited, Mazumdar Shaw multispecialty Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided